CLINICAL TRIAL: NCT05701956
Title: Intravenous Tenecteplase Plus Endovascular Thrombectomy Versus Endovascular Thrombectomy Alone on 4.5 to 24 Hours After Stroke Due to Basilar Artery Occlusion -a Multicenter, Randomized Controlled, Clinical Trial
Brief Title: Intravenous Tenecteplase Plus EVT Versus EVT Alone on 4.5 to 24 Hours After Basilar Artery Occlusion
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: The First Affiliated Hospital of University of Science and Technology of China (Other)
Responsible Party: Principal Investigator, Wei Hu, Professor, The First Affiliated Hospital of University of Science and Technology of China
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ATTENTION LATE
Record Dates: First submitted 2023-01-18; First posted 2023-01-27 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-07

CONDITIONS: Basilar Artery Occlusion; Acute Cerebrovascular Accident; Stroke Due to Basilar Artery Occlusion
Keywords: Thrombectomy; Tenecteplase; Mechanical Thrombectomy
MeSH Terms: conditions — Stroke | interventions — Tenecteplase; TNK-tissue plasminogen activator; Thrombectomy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intravenous tenecteplase+endovascular thrombectomy (Experimental): Patients will receive intravenous tenecteplase (0.25mg/kg, max 25mg) plus endovascular thrombectomy.
  Interventions: Drug: Tenecteplase; Procedure: Endovascular thrombectomy
- Endovascular thrombectomy alone (Active Comparator): Patients will receive endovascular thrombectomy alone.
  Interventions: Procedure: Endovascular thrombectomy

INTERVENTIONS:
Drug: Tenecteplase — Patients will receive intravenous tenecteplase (0.25mg/kg, maximum 25mg, administered as a bolus over 5-10 seconds) before endovascular thrombectomy
  Other Names: TNK; TNK-tPA; TNKase; rhTNK-tPA
  Arms: Intravenous tenecteplase+endovascular thrombectomy
Procedure: Endovascular thrombectomy — The choice of endovascular thrombectomy strategy will be made by the treating neurointerventionist. All thrombectomy devices for endovascular treatment, which are approved by CFDA for this purpose, are allowed in the trial.
  Other Names: thrombectomy

SUMMARY:
To assess the effect of intravenous tenecteplase plus endovascular thrombectomy (EVT) compared to EVT alone on 4.5 to 24 hours after stroke due to basilar artery occlusion.

DETAILED DESCRIPTION:
Background and Rationale: Recently, two prospective multicenter RCT (ATTENTION and BAOCHE trials) have shown a significantly beneficial effect of EVT in patients with an acute symptomatic basilar artery occlusion. The EXTEND-IA TNK trial demonstrated that intravenous thrombolysis with tenecteplase is superior to alteplase before EVT for anterior circulation large vessel occlusion strokes. However, it is unclear whether intravenous tenecteplase bridging with EVT is superior to EVT alone in the extended window patients with basilar artery occlusion. Therefore, additional studies are needed to explore the potential benefit of intravenous tenecteplase in these patients.

Study design: Multicenter, prospective, controlled clinical trial with open-label treatment and blind outcome assessment (PROBE) of intravenous tenecteplase plus EVT versus EVT alone. The trial has observer blinded assessment of the primary outcome and neuroimaging at baseline and follow up.

ELIGIBILITY:
Inclusion Criteria:

1. Patients presenting with posterior circulation ischemic stroke symptoms due to basilar artery occlusion or vertebral artery occlusions that prevent antegrade flow into the basilar artery;
2. Time from stroke onset to randomization within 4.5-24 hours of estimated time of basilar artery occlusion;
3. Patient's age≥18 years;
4. Presence of basilar artery or vertebral artery occlusion, confirmed by CT Angiography (CTA), MR Angiography (MRA) or Digital Subtraction Angiography (DSA). In cases of vertebral artery occlusion, the occlusion must completely prevent antegrade flow into the basilar artery;
5. Patients presenting with acute ischemic stroke eligible using standard criteria (except for time window) to receive both endovascular thrombectomy and intravenous thrombolysis;
6. Baseline National Institutes of Health Stroke Scale (NIHSS) score≥ 10 at the time of neuroimaging;
7. The patient or patient's legal representative signs the informed consent form.

Exclusion Criteria:

1. CT or MR evidence of intracerebral hemorrhage (the presence of < 10 microbleeds is allowed);
2. Pre-stroke modified Rankin scale (mRS) score of ≥ 2;
3. Posterior circulation Acute Stroke Prognosis Early CT Score (PC-ASPECTS) on CT/ CTA-Source Images<6; PC-ASPECTS on magnetic resonance imaging-diffusion weighted imaging (MRI-DWI) <5;
4. Pregnant or lactating women;
5. Allergy to contrast agent or nitinol alloy;
6. Life expectancy<1 year;
7. CTA/MRA/DSA show vascular tortuosity, vascular variation or artery dissection, which would make it difficult to perform endovascular treatment;
8. Participating in other clinical trials;
9. Systolic blood pressure >185 mmHg or diastolic blood pressure >110 mmHg, which cannot be controlled by antihypertensive drugs;
10. Genetic or acquired hemorrhagic diathesis, lack of anticoagulant factor; or oral anticoagulant with international normalized ratio (INR) > 1.7, or novel oral anticoagulant within prior 48 hours;
11. Blood glucose <50 mg/dl (2.8 mmol/L) or >400 mg/dl (22.2 mmol/L), platelet< 100*109/L;
12. Renal insufficiency defined as serum creatinine >2.0 mg/dl (or 176.8 μ mol/l) or a glomerular filtration rate <30 mL/min or the need for hemodialysis or peritoneal dialysis;
13. Patients who cannot complete 90-day follow-up (such as patients without fixed residence, overseas patients, etc);
14. The patient has acute ischemic cerebral infarction within 3 months from randomization;
15. The patient had a history of or clinical suspicion for cerebral vasculitis or infectious endocarditis;
16. The patient has nervous system disease or mental disorder before stroke onset, which may affect the assessment of their condition;
17. CT or MR examination showed large cerebellar infarction with obvious space occupying effect and compression of the fourth ventricle;
18. Patients with extensive bilateral thalamic or extensive bilateral brainstem infarction on CT or MR examination;
19. CTA/MRA/DSA show both anterior and posterior circulation large vessel occlusion;
20. Patients with intracranial tumors (except small meningiomas);
21. Patients who received intravenous thrombolytics treatment before the randomization;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 332 (Estimated)
Dates: Start 2023-03-16 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with modified Rankin Score 0-2 at day 90 (±14 days) | 90 (± 14 days) after procedure
  modified Rankin scale (range, 0 to 6, with a score of 0 indicating no disability, 1 no clinically significant disability, 2 slight disability, 3 moderate disability but remaining able to walk unassisted, 4 moderately severe disability, 5 severe disability, and 6 death)

SECONDARY OUTCOMES:
Proportion of patients with modified Rankin Score 0-3 at day 90 (±14 days) | 90 (± 14 days) after procedure
  modified Rankin scale (range, 0 to 6, with a score of 0 indicating no disability, 1 no clinically significant disability, 2 slight disability, 3 moderate disability but remaining able to walk unassisted, 4 moderately severe disability, 5 severe disability, and 6 death)
Ordinal Shift analysis of modified Rankin Score at day 90 (±14 days) | 90 (± 14 days) after procedure
  modified Rankin scale (range, 0 to 6, with a score of 0 indicating no disability, 1 no clinically significant disability, 2 slight disability, 3 moderate disability but remaining able to walk unassisted, 4 moderately severe disability, 5 severe disability, and 6 death)
Score on the NIHSS at 24 hours | 24 hours after procedure
  The NIHSS is an ordinal hierarchical scale to evaluate the severity of stroke by assessing a patient's performance. Scores range from 0 to 42, with higher scores indicating a more severe deficit.
Score on the NIHSS at 5-7 days or discharge | 5-7 days or discharge after procedure
  The NIHSS is an ordinal hierarchical scale to evaluate the severity of stroke by assessing a patient's performance. Scores range from 0 to 42, with higher scores indicating a more severe deficit.
Proportion of patients with modified Rankin Score 0-1 at day 90 (±14 days) | 90 (± 14 days) after procedure
  modified Rankin scale (range, 0 to 6, with a score of 0 indicating no disability, 1 no clinically significant disability, 2 slight disability, 3 moderate disability but remaining able to walk unassisted, 4 moderately severe disability, 5 severe disability, and 6 death)
Proportion of patients with modified Rankin Score 0-4 at day 90 (±14 days) | 90 (± 14 days) after procedure
  modified Rankin scale (range, 0 to 6, with a score of 0 indicating no disability, 1 no clinically significant disability, 2 slight disability, 3 moderate disability but remaining able to walk unassisted, 4 moderately severe disability, 5 severe disability, and 6 death)
Score on the EuroQoL 5-dimensions 5-level (EQ5D-5L) at 90 days (±14 days) | 90 (± 14 days) after procedure
  Health-related quality of life, assessed with EQ-5D-5L
level of activities of daily living (Barthel index, BI) at 90 days (±14 days) | 90 (± 14 days) after procedure
  Level of activities of daily living
Successful reperfusion (Extended thrombolysis in cerebral infarction [eTICI] score 2b50-3) on digital substraction angiography (DSA) prior to thrombectomy | within 5 minutes at angiography
  Evaluate effect of intravenous thrombolysis on reperfusion
Successful reperfusion on final angiography of thrombectomy | Within 5 minutes at final angiography of thrombectomy
  Evaluate effect of thrombectomy on reperfusion
Successful recanalization on CT or MR angiography within 72 hours | Within 72 hours after procedure
  Evaluate vascular patency after treatment
Infarct volume (Posterior Circulation Acute Stroke Prognosis Early Computed Tomography Score, PC-ASPECTS) evaluated on CT or MRI within 72 hours | Within 72 hours after procedure
  PC-ASPECTS=10 indicates a normal scan, PC-ASPECTS=0 indicates early ischemic changes or hypoattenuation in all above territories. 1 or 2 points each are subtracted for early ischemic changes or hypoattenuation in: left or right thalamus, cerebellum or posterior cerebral artery territory, respectively (1 point); any part of midbrain or pons (2 points)

OTHER OUTCOMES:
Overall mortality at 7 (± 2 days) and 90 (± 14 days) | 7 (± 2 days) and 90 (± 14 days) after procedure
  evaluate death rate
Symptomatic intracerebral hemorrhage (sICH) within 72 hours | Within 72 hours after procedure
  SICH means any hemorrhage with neurological deterioration, as indicated by an NIHSS score that was higher by ≥4 points than the value at baseline or the lowest value in the first 72 hours or any hemorrhage leading to death
Any intracerebral hemorrhage within 72 hours | Within 72 hours after procedure
  Evaluate intracerebral hemorrhage

CONTACTS AND LOCATIONS:
Overall Officials: Wei Hu, MD, Study Chair — The First Affiliated Hospital of University of Science and Technology of China
Locations (1):
- The First Affiliated Hospital of University of Science and Technology of China, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No